CLINICAL TRIAL: NCT01185522
Title: Pharmacoepidemiological Study of the Impact of Roactemra® Treatment on Fatigue in Rheumatoid Arthritis Patients in a Real Life Setting
Brief Title: An Observational Study of the Impact of RoActemra/Actemra on Fatigue in Patients With Rheumatoid Arthritis (PEPS)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22457
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab: Eligible participants receiving tocilizumab according to summary of product characteristics in a real life setting will be observed for 4 months

SUMMARY:
This prospective, observational study will assess the effect of RoActemra/Actemra (tocilizumab) on fatigue in patients with moderate to severe rheumatoid arthritis who have an inadequate response to disease-modifying antirheumatic drugs (DMARDS) or anti tumor necrosis factor (anti-TNF) drugs. Eligible patients receiving RoActemra/Actemra according to the standard of care will be followed for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis
* Inadequate response to disease-modifying antirheumatic drugs (DMARDS) or anti-TNF (tumor necrosis factor) drugs

Exclusion Criteria:

* Hypersensitivity to RoActemra/Actemra or any component
* Active infection
* Participation in a clinical trial in rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inadequate response to DMARDs or anti-TNF receiving RoActemra/Actemra according to standard of care
Sampling Method: Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 719 participants were enrolled in this study conducted from Jan 2010 to May 2011 at 20 centers in France
Pre-assignment Details: Of 719 participants, 25 did not respect inclusion criteria (age less than 18 years or missing age, no or missing attestation of information about the study) and one did not receive any tocilizumab (RoActemra®) infusion.
Groups:
- Tocilizumab: Eligible participants who were receiving tocilizumab according to summary of product characteristics in a real life setting were observed for 4 months.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 693
Completed | 585
Not Completed | 108
Not completed — Lack of Efficacy | 28
Not completed — Lost to Follow-up | 19
Not completed — Withdrawal by Subject | 10
Not completed — Poor tolerance | 39
Not completed — Other reasons | 12

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants included in the study who respected the inclusion and non-inclusion criteria and received at least one tocilizumab infusion.
Groups:
- Tocilizumab: Participants who received tocilizumab according to summary of product characteristics in a real life setting were observed for 4 months.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 693
Age, Continuous [Mean (Standard Deviation); unit: Year] | 55.65 (13.09)
Sex/Gender, Customized [Number; unit: participants]
  Female | 561
  Male | 125
  Missing | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Clinically Significant Improvement in Fatigue After 4 Months of Tocilizumab Treatment
Description: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score assesses self-reported fatigue and its impact upon daily activities and function. It is calculated with 13-item questionnaire on 5-point scale: 0 (not at all) to 4 (very much). The larger the participant's response to the questions (exception of 2 negatively stated), the greater the participants fatigue. For all questions (except for 2 negatively stated), the code is reversed and a new score is calculated as 4 minus the participant's response. The sum of all responses resulted a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status. Clinically relevant improvement is defined as a >= 4-point change from Baseline.
  This was performed using the last observation carried forward (LOCF) method and for participants who completed a FACIT-Fatigue score at Month 4 (completers).
Time Frame: At Month 4
Population: Patient analysis population consisted of all participants included in the study, who respected inclusion criteria, received at least one tocilizumab infusion, had an evaluable FACIT-Fatigue score at inclusion, and at least one evaluable FACIT fatigue score during treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 610
Percentage of participants | 63.3 [58.7 to 67.9]

2. Secondary Outcome: Baseline Disease Characteristics: Mean Disease Duration
Description: Mean disease (rheumatoid arthritis) duration at inclusion was recorded for all participants as baseline disease characteristics.
Time Frame: Baseline (Day [D] 0)
Population: Patient analysis population was considered. Participants for whom data of disease duration was available at baseline were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Tocilizumab
Number analyzed (Participants) | 609
years | 11.7 (9.5)

3. Secondary Outcome: Baseline Disease Characteristics: Number of Participants With Positive Rheumatoid Factor and/or Anti-cyclic Citrullinated Protein Antibodies
Description: Blood was collected for Rheumatoid Factor (RF) at Baseline and was analyzed. RF level was reported in international units/milliliter (IU/mL). All participants were assessed for anti-cyclic citrullinated protein (anti-CCP) antibodies at baseline. Number of participants with a positive RF and/or anti-CCP antibodies were reported as baseline disease characteristics.
Time Frame: Baseline (D0)
Population: Patient analysis population was considered. Participants with positive RF and/or anti-CCP antibodies at baseline were analyzed for this outcome measure.
Measure: Number; unit: Number of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 572
Number of Participants | 463

4. Secondary Outcome: Baseline Disease Characteristics: Tender Joint Count and Swollen Joint Count
Description: For tender joint count, a total of 68 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no tender joint) to 68 (worse possible score or all tender joints). Lower scores indicate no tender joint and higher scores indicate worsening tender joints.
  For swollen joint count, a total of 66 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no swollen joint) to 66 (worse possible score or all swollen joints). Lower scores indicate no swollen joint and higher scores indicate worsening swollen joints. Tender joint count and swollen joint count were assessed at baseline and were used as baseline disease characteristics for assessment of rheumatoid arthritis.
Time Frame: Baseline (D0)
Population: Patient analysis population was considered. n = number of participants available for particular parameters.
Measure: Mean (Standard Deviation); unit: Number of joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 606
Number of joints
  TJC (n = 606) | 9.9 (6.6)
  SJC (n = 605) | 6.6 (5.1)

5. Secondary Outcome: Baseline Disease Characteristic: DAS28, Patient's Global Assessment, VAS Pain and HAQ Score as Rheumatoid Arthritis Assessment Parameters
Description: DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/h), and patient's global assessment of disease activity (measured on a 100-mm visual analog scale, where 0 is no disease activity and 100 is maximum disease activity). The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening disease activity. VAS pain score calculated as 0 to 10 cm; where 0 = no pain, and 10 = worst possible pain. HAQ indicates how the disease affected participant's activities of daily life. It consisted of 20 questions in 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale, 0=without any difficulty to 3=unable to do. Sum of scores was divided by number of domains with a score for a total possible score of 0 (best/no difficulties to perform activities) to 3 (worst/ unable to perform activities at all).
Time Frame: Baseline (D0)
Population: Patient analysis population consisted of all participants included in the study, who respected inclusion criteria, received at least one tocilizumab infusion, had an evaluable FACIT-Fatigue score at inclusion, and at least one evaluable FACIT fatigue score during treatment. n = number of participants available for particular parameters.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 608
Scores on a scale
  DAS28 (n = 563) | 5.3 (1.1)
  Patient's global assessment (VAS) (n = 594) | 63.9 (22.0)
  VAS Pain (n = 597) | 62.7 (22.8)
  HAQ score (n = 608) | 1.6 (0.7)

6. Secondary Outcome: Baseline Disease Characteristic: Number of Participants With High Erythrocyte Sedimentation Rate, CRP Level, Anemia, and Unacceptable Patient Acceptable Symptom State Fatigue
Description: High Erythrocyte Sedimentation Rate (ESR) was defined as (1) for participants aged up to 50 years: > 15 mm/h for men and > 20 mm/h for women, and (2) for participants aged over 50 years: > 20 mm/h for men and > 25 mm/h for women. Anemia was defined as plasma hemoglobin level <12 gram per deciliter (g/dL) for women and <13 g/dL for men. The CRP test is evaluated for an acute phase reactant of inflammation. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Patient-Acceptable Symptom State (PASS) that is defined as the highest level of symptom beyond which participants consider themselves well. PASS is a 1-question assessment of how rheumatoid arthritis has affected participant in last 48 hours.
Time Frame: Baseline (D0)
Population: as for outcome 5
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 595
Number of participants
  High ESR (n = 577) | 307
  CRP > 10 mg/L (n = 595) | 278
  Anemia (n = 574) | 148
  Unacceptable PASS fatigue (n = 578) | 423

7. Secondary Outcome: Baseline Disease Characteristic: Mean FACIT-Fatigue Score and VAS Fatigue Score
Description: FACIT-fatigue score and VAS fatigue score were fatigue assessment parameters. FACIT-Fatigue score assesses self-reported fatigue and its impact upon daily activities and function. It is calculated with 13-item questionnaire on 5-point scale, 0 (not at all) to 4 (very much). The larger the participant's response to the questions (exception of 2 negatively stated), the greater the participants fatigue. For all questions (except for 2 negatively stated), the code is reversed and a new score is calculated as 4 minus the participant's response. The sum of all responses results a total possible score of 0 (worse score) to 52 (better score). VAS fatigue score ranges from 0 (symptom-free and no arthritis symptoms) to 100 (worsening in symptoms and arthritis disease activity). Clinically relevant improvement is defined as >/= 4-point change from Baseline.
Time Frame: Baseline (D0)
Population: Patient analysis population consisted of all participants included in the study, who respected inclusion criteria, received at least one tocilizumab infusion, had an evaluable FACIT-Fatigue score at inclusion, and at least one evaluable FACIT fatigue score during treatment. n = number of participants available for particular time fatigue scores.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 610
Scores on a scale
  FACIT-Fatigue score (n = 610 ) | 24.4 (10.5)
  VAS Fatigue (n = 602) | 61.3 (23.2)

8. Primary Outcome: Number of Participants With Clinically Significant Improvement in Fatigue at Month 4 With Respect to Predictive Factors
Description: Predictive factors of fatigue were taken into account included gender, age, time since initial diagnosis, Erosive RA, disease activity score (DAS, ranging from 0 [no disease activity] to 10 [worsening in disease activity]), erythrocyte sedimentation rate (ESR), anemia, treatment with corticosteroids, doses of corticosteroids, health assessment questionnaire (HAQ, ranging from 0 [without any difficulty] to 60 [worsening or unable to do physical activities]), FACIT-Fatigue score (ranging from 0 [worse score] to 52 [better score]), visual analogue score (VAS) for fatigue, pain, quality of sleep, and global assessment (ranging from 0 [symptom-free and no arthritis symptoms] to 100 [worsening of symptoms and arthritis disease activity]), Short Form 36 (SF36) vitality score (ranging from 0 [worst] to 100 [best]), Hospital Anxiety and Depression Scale (HADS; represented as score </= 7 [no case], 7 to 10 [doubtful case], and > 10 [certain case of HAD]).
Time Frame: At Month 4
Population: Patient analysis population was considered. Participants whom baseline characteristics were available at inclusion and who completed a FACIT-Fatigue score at Month 4 and had clinically significant improvement in fatigue with respect to predictive factors were analyzed for this outcome measure.
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 264
Number of participants
  Gender- female | 214
  Gender- male | 46
  Gender - missing | 4
  Age (<= 55 years) | 139
  Age (> 55 years) | 125
  Time since initial diagnosis (>= 10 years) | 108
  Time since initial diagnosis (< 10 years) | 155
  Erosive RA | 187
  DAS-28 (<= 5.1) | 87
  DAS-28 (> 5.1) | 158
  ESR (<= 28 mm/h) | 134
  ESR (> 28 mm/h) | 118
  Anemia | 69
  Corticosteroids treatment | 178
  HAQ score (<= 1.5) | 118
  HAQ score (> 1.5) | 146
  VAS patient: fatigue (<= 66) | 115
  VAS patient: fatigue (> 66) | 146
  VAS patient: pain (<= 66) | 109
  VAS patient: pain (> 66) | 150
  VAS patient: quality of sleep (<= 30) | 62
  VAS patient: quality of sleep (30 to 59) | 60
  VAS patient: quality of sleep (59 to 77) (n=264) | 60
  VAS patient: quality of sleep (> 77) (n=264) | 76
  VAS patient: global assessment (<= 67) | 112
  VAS patient: global assessment (> 67) | 146
  SF36 vitality score (> 33) | 107
  SF36 vitality score (<= 33) | 145
  HADS score: Anxiety (No case) | 80
  HADS score: Anxiety (Doubtful case) | 61
  HADS score: Anxiety (Certain case) | 103
  HADS score: Depression (No case) | 114
  HADS score: Depression (Doubtful case) | 69
  HADS score: Depression (Certain case) | 69
Statistical Analysis 1: Comparison: Tocilizumab; Comparison between genders: women and men; Test type: Superiority or Other; p = 0.235, Univariate logistic regression model; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.45 to 1.22]
Statistical Analysis 2: Comparison: Tocilizumab; Comparison between Age: <= 55 years and > 55 years; Test type: Superiority or Other; p = 0.331, Univariate logistic regression model; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.55 to 1.22]
Statistical Analysis 3: Comparison: Tocilizumab; Comparison between time since initial diagnosis: >= 10 years and < 10 years; Test type: Superiority or Other; p = 0.050, Univariate logistic regression model; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.00 to 2.23]
Statistical Analysis 4: Comparison: Tocilizumab; Comparison between participants without erosive rheumatoid arthritis (RA) and participants with erosive RA; Test type: Superiority or Other; p = 0.144, Univariate logistic regression model; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.88 to 2.46]
Statistical Analysis 5: Comparison: Tocilizumab; Comparison between DAS-28 score: <= 5.1 and DAS-28 >5.1; Test type: Superiority or Other; p = 0.010, Univariate logistic regression model; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.14 to 2.65]
Statistical Analysis 6: Comparison: Tocilizumab; Comparison between ESR: <= 28 mm/h and > 28 mm/h; Test type: Superiority or Other; p = 0.119, Univariate logistic regression model; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.92 to 2.10]
Statistical Analysis 7: Comparison: Tocilizumab; Comparison between number of participants without anemia and number of participants with anemia; Test type: Superiority or Other; p = 0.265, Univariate logistic regression model; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.81 to 2.13]
Statistical Analysis 8: Comparison: Tocilizumab; Comparison between dose of corticosteroids: <= 5 mg and > 5 mg; Test type: Superiority or Other; p = 0.511, Univariate logistic regression model; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.77 to 1.71]
Statistical Analysis 9: Comparison: Tocilizumab; Comparison between HAQ score: <= 1.5 and > 1.5; Test type: Superiority or Other; p = 0.153, Univariate logistic regression model; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.90 to 2.00]
Statistical Analysis 10: Comparison: Tocilizumab; Comparison between VAS patient: fatigue <= 66 and > 66; Test type: Superiority or Other; p < 0.001, Univariate logistic regression model; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.45 to 3.31]
Statistical Analysis 11: Comparison: Tocilizumab; Comparison between VAS patient: pain <= 66 and > 66; Test type: Superiority or Other; p < 0.001, Univariate logistic regression model; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.35 to 3.08]
Statistical Analysis 12: Comparison: Tocilizumab; Comparison between VAS patient (quality of sleep) score: <=30 score and 30 - 59 score; Test type: Superiority or Other; p = 0.261, Univariate logistic regression model; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.86 to 2.75]
Statistical Analysis 13: Comparison: Tocilizumab; Comparison between VAS patient (quality of sleep) score: <= 30 and 59 - 77; Test type: Superiority or Other; p = 0.261, Univariate logistic regression model; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.67 to 2.05]
Statistical Analysis 14: Comparison: Tocilizumab; Comparison between VAS patient (quality of sleep) score: <= 30 and > 77; Test type: Superiority or Other; p = 0.261, Univariate logistic regression model; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.95 to 2.89]
Statistical Analysis 15: Comparison: Tocilizumab; Comparison between VAS patient: global assessment score: <= 67 and > 67; Test type: Superiority or Other; p < 0.001, Univariate logistic regression model; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.38 to 3.14]
Statistical Analysis 16: Comparison: Tocilizumab; Comparison between SF36 vitality score: > 33 and <= 33; Test type: Superiority or Other; p < 0.001, Univariate logistic regression model; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.50 to 3.47]
Statistical Analysis 17: Comparison: Tocilizumab; Comparison between HADS score: Anxiety (No case) and HADS score: Anxiety (Doubtful case); Test type: Superiority or Other; p = 0.399, Univariate logistic regression model; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.60 to 1.93]
Statistical Analysis 18: Comparison: Tocilizumab; Comparison between HADS score: Anxiety (No case) and HADS score: Anxiety (Certain case); Test type: Superiority or Other; p = 0.399, Univariate logistic regression model; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.48 to 1.26]
Statistical Analysis 19: Comparison: Tocilizumab; Comparison between HADS score: Depression (No Case) and HADS score: Depression (Doubtful case); Test type: Superiority or Other; p = 0.858, Univariate logistic regression model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.65 to 1.81]
Statistical Analysis 20: Comparison: Tocilizumab; Comparison between HADS score: Depression (No Case) and HADS score: Depression (Certain case); Test type: Superiority or Other; p = 0.858, Univariate logistic regression model; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.57 to 1.52]
Statistical Analysis 21: Comparison: Tocilizumab; Comparison between time since initial diagnosis: >= 10 years and < 10 years; Test type: Superiority or Other; p = 0.036, Multivariate logistic regression model; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.03 to 2.58]

9. Primary Outcome: Median Clinically Significant Improvement in C-Reactive Protein as a Predictive Factors After 4 Months of Tocilizumab Treatment
Description: Predictive factors were characteristics of participants that indicated greater or lesser likelihood of responding to a specific treatment regimen. C-reactive protein (CRP) is one of the biomarkers for the diagnosis and assessment of disease activity in RA.
Time Frame: At Month 4
Population: Patient analysis population was considered. Participants who completed a FACIT-Fatigue score at Month 4 and had clinically significant improvement in fatigue with respect to predictive factors were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: milligram per liter
Arm/Group | Tocilizumab
Number analyzed (Participants) | 264
milligram per liter | 13.0 [5.0 to 32.3]
Statistical Analysis 1: Comparison: Tocilizumab; Predictive factor: C-Reactive Protein; Test type: Superiority or Other; p = 0.004, Univariate logistic regression model; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.05 to 1.28]
Statistical Analysis 2: Comparison: Tocilizumab; Predictive factor: C-Reactive Protein; Test type: Superiority or Other; p = 0.013, Multivariate logistic regression model; Odds Ratio (OR) = 1.14, 95% CI 2-sided [1.03 to 1.27]

10. Primary Outcome: Mean Clinically Significant Improvement in Tender Joints and Swollen Joints as Predictive Factors After 4 Months of Tocilizumab Treatment
Description: Predictive factors were characteristics of participants that indicated greater or lesser likelihood of responding to a specific treatment regimen.
  For tender joint count (TJC), a total of 68 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no tender joint) to 68 (worse possible score or all tender joints). Lower scores indicate no tender joint and higher scores indicate worsening tender joints.
  For swollen joint count (SJC), a total of 66 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no swollen joint) to 66 (worse possible score or all swollen joints). Lower scores indicate no swollen joint and higher scores indicate worsening swollen joints.
Time Frame: At Month 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Number of joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 264
Number of joints
  Number of tender joints | 10.02 (6.72)
  Number of swollen joints | 7.28 (5.36)
Statistical Analysis 1: Comparison: Tocilizumab; Predictive factor: Tender joint; Test type: Superiority or Other; p = 0.253, Univariate logistic regression model; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.99 to 1.05]
Statistical Analysis 2: Comparison: Tocilizumab; Predictive factor : Swollen joint; Test type: Superiority or Other; p = 0.021, Univariate logistic regression model; Odds Ratio (OR) = 1.05, 95% CI 2-sided [1.01 to 1.09]

11. Secondary Outcome: Correlation Between Relative Changes From Baseline of FACIT-Fatigue Score and VAS Fatigue to 4 Months of Tocilizumab Treatment
Description: Correlation between FACIT-Fatigue score and VAS fatigue was evaluated for all participants at inclusion and after 4 months of tocilizumab treatment (relative change from baseline) using a linear regression. FACIT-Fatigue score assesses self-reported fatigue and its impact upon daily activities and function. It is calculated with 13-item questionnaire on 5-point scale, 0 (not at all) to 4 (very much). The larger the participant's response to the questions (exception of 2 negatively stated), the greater the participants fatigue. For all questions (except for 2 negatively stated), the code is reversed and a new score is calculated as 4 minus the participant's response. The sum of all responses results a total possible score of 0 (worse score) to 52 (better score). VAS fatigue score ranging from 0 (symptom-free and no arthritis symptoms) to 100 (worsening in symptoms and arthritis disease activity)
Time Frame: From Baseline (D0) to Month (M) 4
Population: Patient analysis population was considered. Participants with Changes in FACIT-Fatigue Score and VAS Fatigue at Month 4 were analyzed for this outcome measure.
Measure: Number; unit: Correlation Coefficient
Arm/Group | Tocilizumab
Number analyzed (Participants) | 87
Correlation Coefficient | -0.1736

12. Secondary Outcome: Median Time to Onset of an Improvement of the FACIT-Fatigue Score
Description: The time of onset of a clinically significant improvement of fatigue was defined as the time between the date of the first tocilizumab infusion and the date of the first increase of at least 4 points of the FACIT-Fatigue score (date of questionnaire completion) during 4 months of tocilizumab treatment. FACIT-Fatigue score assesses self-reported fatigue and its impact upon daily activities and function. It is calculated with 13-item questionnaire on 5-point scale, 0 (not at all) to 4 (very much). The larger the participant's response to the questions (exception of 2 negatively stated), the greater the participants fatigue. For all questions (except for 2 negatively stated), the code is reversed and a new score is calculated as 4 minus the participant's response. The sum of all responses results a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Up to Month 4
Population: Patient analysis population was considered. Participants with increase of at least 4 points of the FACIT-Fatigue score were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tocilizumab
Number analyzed (Participants) | 264
Months | 1.0 [1.0 to 1.3]

13. Secondary Outcome: Relative Median Change From Baseline in DAS 28 and VAS Patient's Global Assessment to Month 1, Month 2, Month 3, and Month 4
Description: Relative change from Baseline (BL) in DAS 28 was evaluated for all participants at each evaluation time (on raw data at inclusion; at Month 1, Month 2, Month 3, and Month 4 using a linear regression. DAS-28 and VAS patient's global assessment (PGA) were described as continuous variables for all participants at each evaluation time points (Baseline to M4). DAS 28 ranging from 0 (no disease activity) to 10 (worsening in disease activity) and VAS PGA ranging from 0 (symptom-free and no arthritis symptoms) to 100 (worsening of symptoms and arthritis disease activity),
Time Frame: From Baseline (D0) to M 1, M 2, M 3, and M 4
Population: Patient analysis population was considered. Participants with changes in DAS 28 up to Month 4 were analyzed for this outcome measure. n = number of participants available for particular parameters at specified time points.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 519
Percent change
  Change from BL in DAS28 to M1 (n=462) | -30.9 [-84.0 to 71.0]
  Change from BL in DAS-28 at M2 (n=431) | -40.5 [-91.5 to 45.8]
  Change from BL in DAS-28 at M3 (n=416) | -46.1 [-92.3 to 89.9]
  Change from BL in DAS-28 at M4 (n=366) | -48.4 [-98.8 to 62.7]
  Change from BL in VAS PGA at M1 (n=519) | -21.7 [-100.0 to 700.0]
  Change from BL in VAS PGA at M2 (n=477) | -34.8 [-100.0 to 1040.0]
  Change from BL in VAS PGA at M3 (n=460) | -40.0 [-100.0 to 1060.0]
  Change from BL in VAS PGA at M4 (n=405) | -42.9 [-100.0 to 376.2]

14. Secondary Outcome: Relative Median Change From Baseline in Disease Activity (Tender Joint Count and Swollen Joint Count) to Month 1, Month 2, Month 3, and Month 4
Description: Relative change (RC) from Baseline (BL) in disease activity included TJC and SJC was evaluated as continuous variables for all participants at each evaluation time points.
  For tender joint count, a total of 68 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no tender joint) to 68 (worse possible score or all tender joints). Lower scores indicate no tender joint and higher scores indicate worsening tender joints. For swollen joint count, a total of 66 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no swollen joint) to 66 (worse possible score or all swollen joints). Lower scores indicate no swollen joint and higher scores indicate worsening swollen joints.
Time Frame: From Baseline (D0) to M 1, M 2, M 3, and M 4
Population: Patient analysis population was considered. Participants with changes in TJC and SJC up to Month 4 were analyzed for this outcome measure. n = number of participants available for particular parameters at specified time points.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 578
Percent change
  RC from BL of TJC at M1 (n=578) | -34.3 [-100.0 to 1600.0]
  RC from BL of TJC at M2 (n=558) | -55.3 [-100.0 to 950.0]
  RC from BL of TJC at M3 (n=537) | -66.7 [-100.0 to 550.0]
  RC from BL of TJC at M4 (n=498) | -67.3 [-100.0 to 1200.0]
  RC from BL of SJC at M1 (n=546) | -42.9 [-100.0 to 1100.0]
  RC from BL of SJC at M2 (n=530) | -60.0 [-100.0 to 1300.0]
  RC from BL of SJC at M3 (n=507) | -69.2 [-100.0 to 700.0]
  RC from BL of SJC at M4 (n=470) | -75.0 [-100.0 to 700.0]

15. Secondary Outcome: Relative Median Change From Baseline in ESR to Month 1, Month 2, Month 3, and Month 4
Description: The correlation between fatigue and ESR value was evaluated for all participants at each evaluation time (on raw data at inclusion; on relative changes at M1 to M4) using a linear regression. ESR values were described as continuous variables for all participants at each evaluation time (Baseline to M4).
Time Frame: From Baseline (D0) to M 1, M 2, M 3, and M 4
Population: Patient analysis population was considered. Participants with Changes in ESR values up to Month 4 were analyzed for this outcome measure. n = number of participants available at specified time points.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 537
Percent change
  M1 (n=537) | -70.0 [-97.9 to 860.0]
  M2 (n=530) | -75.0 [-98.8 to 600.0]
  M3 (n=514) | -78.1 [-98.9 to 385.7]
  M4 (n=476) | -78.6 [-100.0 to 1450.0]

16. Secondary Outcome: Relative Median Change From Baseline in C - Reacting Protein at Month 1, Month 2, Month 3, and Month 4
Description: The correlation between fatigue and CRP value was evaluated for all participants at each evaluation time (on raw data at inclusion; on relative changes at M1 to M4) using a linear regression. CRP values were described as continuous variables for all participants at each evaluation time (Baseline to M4).
Time Frame: From Baseline (D0) to M 1, M 2, M 3, and M 4
Population: Patient analysis population was considered. Participants with Changes in CRP level up to Month 4 were analyzed for this outcome measure. n = number of participants available at specified time points.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 561
Percent change
  M1 (n=561) | -76.6 [-100.0 to 1600.0]
  M2 (n=549) | -80.0 [-100.0 to 1080.0]
  M3 (n=531) | -80.4 [-100.0 to 1005.3]
  M4 (n=493) | -81.3 [-100.0 to 2400.0]

17. Secondary Outcome: Number of Participants Achieving PASS Score at Baseline (Day 0) and Month 4
Description: A PASS score at Day 0 and Month 4 calculated on participants with acceptable symptom state. PASS is defined as the highest level of symptom beyond which participants consider themselves well. PASS is a 1-question assessment of how rheumatoid arthritis has affected participant in last 48 hours.
Time Frame: Baseline (D0) and Month 4
Population: Patient analysis population consisted of all participants included in the study, who respected inclusion criteria, received at least one tocilizumab infusion, had an evaluable FACIT-Fatigue score at inclusion, and at least one evaluable FACIT fatigue score during treatment. n = number of participants available at the particular time point.
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 578
Number of participants
  D0 (n=578) | 155
  M4 (n=403) | 269

18. Secondary Outcome: Percentage of Participants With FACIT-Fatigue Score, SF36 Vitality Score, and VAS Fatigue at Day 0 and Month 4
Description: FACIT-Fatigue score (ranging from 0 [worse score] to 52 [better score]), VAS (ranging from 0 [symptom-free and no arthritis symptoms] to 100 [worsening in arthritis disease activity]) and SF36 vitality score (ranging from 0 [worst] to 100 [best]) were calculated at Baseline and Month 4.
Time Frame: Baseline (D0) and Month 4
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 610
Percentage of participants
  FACIT-Fatigue score at D0 | 39.0
  FACIT-Fatigue score at M4 | 45.0
  SF36 vitality score at D0 | 55.0
  SF36 vitality score at M4 | 60.0
  VAS fatigue at D0 | 61.0
  VAS fatigue at M4 | 47.0

19. Secondary Outcome: Correlations Between Fatigue and Other Participant Reported Outcomes at Day 0 and Month 4
Description: Fatigue was assessed by FACIT-Fatigue scale (ranging from 0 [worse score] to 52 [better score]) and VAS fatigue (ranging from 0 [symptom-free and no arthritis symptoms] to 100 [worsening of symptoms and arthritis disease activity]). Other participant reported outcomes (PROs) were VAS for pain and quality of sleep (ranging from 0 [symptom-free and no arthritis symptoms] to 100 [worsening in arthritis disease activity]), SF36 vitality score (ranging from 0 [worst] to 100 [best]) and HAD score (calculated using the 14 items and each item was scored 0, 1, 2 or 3 where a score of 3 corresponds to the most anxious/depressed. 7-item depression and 7-item anxiety subscales were summed; each resulting in a total score of 0-21). Correlation between fatigue as assessed by FACIT-Fatigue score or VAS fatigue was evaluated for all participants using a linear regression and were reported for D0 and M4.
Time Frame: Day 0 and Month 4
Population: as for outcome 17
Measure: Number; unit: Coefficient of correlation
Arm/Group | Tocilizumab
Number analyzed (Participants) | 610
Coefficient of correlation
  FACIT-Fatigue : VAS pain at D0 | -0.4843
  FACIT-Fatigue : VAS pain at M4 | -0.0656
  FACIT-Fatigue : VAS quality of sleep at D0 | -0.4785
  FACIT-Fatigue : VAS quality of sleep at M4 | -0.1339
  FACIT-Fatigue : SF36 vitality at D0 | 0.7536
  FACIT-Fatigue : SF36 vitality at M4 | 0.6720
  FACIT-Fatigue : HAQ score at D0 | -0.5314
  FACIT-Fatigue : HAQ score at M4 | -0.2248
  FACIT-Fatigue : HADS Anxiety score at D0 | -0.4400
  FACIT-Fatigue : HADS Anxiety score at M4 | -0.1584
  FACIT-Fatigue : HADS Depression score at D0 | -0.5791
  FACIT-Fatigue : HADS Depression score at M4 | -0.2817
  VAS fatigue : VAS pain at D0 | 0.6040
  VAS fatigue : VAS pain at M4 | 0.0273
  VAS fatigue : VAS quality of sleep at D0 | 0.4778
  VAS fatigue : VAS quality of sleep at M4 | 0.0708
  VAS fatigue : SF36 vitality at D0 | -0.5741
  VAS fatigue : SF36 vitality at M4 | -0.1268
  VAS fatigue : HAQ score at D0 | 0.3156
  VAS fatigue : HAQ score at M4 | 0.1320
  VAS fatigue : HADS Anxiety score at D0 | 0.2588
  VAS fatigue : HADS Anxiety score at M4 | -0.0186
  VAS fatigue : HADS Depression score at D0 | 0.3278
  VAS fatigue : HADS Depression score at M4 | 0.0825

20. Secondary Outcome: Number of Participants for Rheumatoid Arthritis Management With Tocilizumab Treatment up to Month 4
Description: Participants with tocilizumab treatment were managed according to number of tocilizumab treatment received according to Summary of Product Characteristics recommendations, as 8 mg/kg, dose duration of 1-hour, correct infusion progress; and received DMARD, methotrexate, and corticosteroids concomitantly with tocilizumab during Months 1 to 4.
Time Frame: From Baseline (D0) to M 1, M 2, M 3, and M 4
Population: as for outcome 17
Measure: Number; unit: Number of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 592
Number of Participants
  Dose 8 mg/kg dose, M1 (n = 590) | 558
  Dose 8 mg/kg dose, M2 (n = 575) | 540
  Dose 8 mg/kg dose, M3 (n = 548) | 511
  Dose 8 mg/kg dose, M4 (n = 512) | 477
  Dose duration 60 minutes, M1 (n = 559) | 472
  Dose duration 60 minutes, M2 (n = 547) | 463
  Dose duration 60 minutes, M3 (n = 516) | 433
  Dose duration 60 minutes, M4 (n = 494) | 426
  Correct infusion progress, M1 (n = 527) | 520
  Correct infusion progress, M2 (n = 516) | 510
  Correct infusion progress, M3 (n = 485) | 482
  Correct infusion progress, M4 (n = 447) | 442
  Concomitant DMARD, M1 (n = 591) | 389
  Concomitant DMARD, M2 (n = 577) | 381
  Concomitant DMARD, M3 (n = 549) | 359
  Concomitant DMARD, M4 (n = 512) | 338
  Concomitant Methotrexate, M1 (n = 591) | 346
  Concomitant Methotrexate, M2 (n = 577) | 341
  Concomitant Methotrexate, M3 (n = 549) | 325
  Concomitant Methotrexate, M4 (n = 512) | 306
  Concomitant corticosteroids, M1 (n = 592) | 391
  Concomitant corticosteroids, M2 (n = 577) | 379
  Concomitant corticosteroids, M3 (n = 549) | 349
  Concomitant corticosteroids, M4 (n = 512) | 320

21. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An Any Adverse Events (AEs) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An Serious Adverse Events (SAEs) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 4 months
Population: Safety population consisted of all participants included in the study, who respected the inclusion and non-inclusion criteria and who at least one tocilizumab infusion.
Measure: Number; unit: Number of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 693
Number of Participants
  Any AEs | 272
  Any SAEs | 27

ADVERSE EVENTS:
Time Frame: Up to Month 4
Description: Adverse event is reported for safety population which consist of all participants who received at least one tocilizumab infusion.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 27/693
Other Adverse Events (participants affected / at risk) | 117/693
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=693)
Arthritis bacterial (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Subdiaphragmatic abscess (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Meniscus removal (Surgical and medical procedures) | 1
Vascular operation (Surgical and medical procedures) | 1
Arteriospasm coronary (Cardiac disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1 — General Disorders and Administration Site Conditions
Hypersensitivity (Immune system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=693)
Bronchitis (Infections and infestations) | 18
Aphthous stomatitis (Gastrointestinal disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 16
Asthenia (General disorders) | 19 — General disorders and administration site conduction
Headache (Nervous system disorders) | 28
Neutropenia (Blood and lymphatic system disorders) | 23
Cytolytic hepatitis (Hepatobiliary disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.